CLINICAL TRIAL: NCT05874336
Title: An Open-Label, Two-Part Study Designed to Assess the Absolute Bioavailability of Aramchol and to Determine the Mass Balance Recovery, Metabolite Profile and Metabolite Identification to Healthy Male Subjects
Brief Title: An Open-Label, Two-Part Study Designed to Assess the Absolute Bioavailability and Mass Balance of Aramchol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galmed Pharmaceuticals Ltd (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aramchol-020
Record Dates: First submitted 2023-04-24; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: NASH
MeSH Terms: interventions — aramchol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose administration of Aramchol in Part 1 and Part 2 (Experimental): 6 subjects received Aramchol in Part 1 and Part 2 of the study
  Interventions: Drug: Aramchol

INTERVENTIONS:
Drug: Aramchol — Aramchol free acid (3β-arachidylamido-7α,12α-dihydroxy-5β-cholan-24-oic acid) is a synthetic small molecule, produced by conjugation of cholic acid (bile acid) and arachidic acid (saturated fatty acid) linked by a stable amide bond.
  Other Names: Aramchol free acid (3β-arachidylamido-7α,12α-dihydroxy-5β-cholan-24-oic acid)

SUMMARY:
A two-part open-label study to assess the absolute bioavailability of aramchol and the mass balance recovery, metabolite profile and identification of metabolite structures for [14C]-aramchol in healthy male subjects

DETAILED DESCRIPTION:
A two-part open-label study to assess the absolute bioavailability of aramchol and the mass balance recovery, metabolite profile and identification of metabolite structures for [14C]-aramchol in healthy male subjects.

A subject was considered evaluable in Part 1 if they provided PK samples for up to a minimum of 120 h after first investigational medicinal product (IMP) administration. A subject was considered evaluable in Part 2 if they provided biological samples for up to a minimum of 144 h after IMP administration or demonstrated >90% mass balance recovery, or <1% of the administered dose eliminated in excreta for 2 consecutive days, whichever was sooner.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Aged 35 to 64 years at the time of signing informed consent
3. Body mass index (BMI) of 18.0 to 35.0 kg/m2 as measured at screening
4. Must be willing and able to communicate and participate in the whole study
5. Must have regular bowel movements (ie average stool production of ≥1 and ≤3 stools per day)
6. Must provide written informed consent
7. Must agree to adhere to the contraception requirements

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. History of any drug or alcohol abuse in the past 2 years
4. Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
5. A confirmed positive alcohol breath test at screening or each admission
6. Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or each admission
7. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
8. Subjects with pregnant or lactating partners
9. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
10. Participation in any study involving administration of any [14C]-labelled compound within 12 months prior to dosing in Part 1 of this study

Ages: 35 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male subjects
Enrollment: 6 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability | 10 days
  Measure the AUC(0-inf) of orally and intravenously (IV) administered Aramchol
Mass balance recovery | 10 days
  Assess the mass balance recovery of total amounts of radioactivity excreted in urine and feces
Metabolite profiling | 10 days
  Assess the potential metabolites of Aramchol and determine their chemical structure in plasma, urine and fecal samples

SECONDARY OUTCOMES:
Routes and rates of elimination | 10 days
  Determine the routes and rates of elimination of [14C]-Aramchol in excreta
Chemical structure of each metabolite accounting for more than 10% | 10 days
  Identify the chemical structure of each metabolite accounting for more than 10% by area under the curve (AUC) of circulating total radioactivity or 10% of the dose in urine and feces
PK- Area under the concentration-time curve (AUC) | 10 days
  Investigate the plasma Area under the concentration-time curve (AUC) of Aramchol
PK- Time of maximum observed concentration (Tmax) | 10 days
  Investigate the plasma Time of maximum observed concentration (Tmax) of Aramchol
PK- Maximum observed concentration (Cmax) | 10 days
  Investigate the plasma Maximum observed concentration (Cmax) of Aramchol
PK- Total body clearance (CL) | 10 days
  Investigate the Total body clearance (CL) of Aramchol
Safety- Adverse events | 10 days
  Assess and characterize the number of participants with adverse events
Safety- Clinical laboratory parameters | 10 days
  Assess and characterize the number of participants with clinically significant changes in clinical laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: John Posner, PhD, FRCP, Study Director — Consultant
Locations (1):
- Quotient Sciences, Mere Way, Ruddington Fields, Ruddington, Nottingham, NG11 6JS, UK., Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Consideration will be made whether to share any data of this mass balance study